CLINICAL TRIAL: NCT04038892
Title: The Effect of Different Virtual Reality-Based Exercise Trainings on Pulmonary Function, Respiratory and Peripheral Muscle Strength, Functional Capacity and Balance in Children With Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Hikmet Uçgun, Research Assistant, PT, PhD (c), Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: bvuhucgun01
Record Dates: First submitted 2019-07-27; First posted 2019-07-31 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Virtual Reality; Exercise Training; Pulmonary Function; Functional Capacity; 6 Minute Walk Test; Balance; Muscle Strength
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Patients in this group will receive conventional chest physiotherapy, two times a day, 7 days a week for 8 weeks. After the training given by the physiotherapist, all exercise sessions will be performed at home.
  Interventions: Other: Conventional Chest Physiotherapy
- Nintendo Wii Fit Training Group (Experimental): In addition to conventional chest physiotherapy programme, patients in this group will also receive Nintendo Wii Fit based exercise training for 40 minutes, 2 times in a week for 8 weeks. All exercise sessions will be supervised by physiotherapist in a clinic per week.
  Interventions: Other: Conventional Chest Physiotherapy; Other: Nintendo Wii Fit Based Exercise Training
- BreathingLabs Breathing Games Training Group (Experimental): In addition to conventional chest physiotherapy programme, patients in this group will also receive BreathingLabs Breathing Games based exercise training for 40 minutes, 2 times in a week for 8 weeks. All exercise sessions will be supervised by physiotherapist in a clinic per week.
  Interventions: Other: Conventional Chest Physiotherapy; Other: BreathingLabs Breathing Games Based Exercise Training

INTERVENTIONS:
Other: Conventional Chest Physiotherapy — Programme will include diaphragmatic breathing exercise, thoracic expansion exercises, incentive spirometer exercise (Triflo), oscillatory PEP (Flutter), postural drainage, coughing techniques and teaching respiratory control.
Other: Nintendo Wii Fit Based Exercise Training — Nintendo Wii Fit based exercise training will be given under the supervision of a physiotherapist. The one session will be included: warm-up exercises for 5 minutes (yoga games; deep breathing and half moon etc.), aerobic exercises for 30 minutes (aerobic games; Twisting and Squat, Step Plus, Jogging Plus and Hula Hoop etc.) and cooling exercises in 5 minutes (yoga games; deep breathing and half moon etc.).
  Arms: Nintendo Wii Fit Training Group
Other: BreathingLabs Breathing Games Based Exercise Training — BreathingLabs Breathing Games based exercise training will be given under the supervision of a physiotherapist. The one session will be included: warm-up exercises for 5 minutes (respiratory control exerice and coughing techniques), breathing games exercises for 30 minutes (breathing games; Kite, Balloon, Pluto, Butterflies and Plane etc.) and cooling exercises in 5 minutes (respiratory control exerice and coughing techniques).
  Arms: BreathingLabs Breathing Games Training Group

SUMMARY:
Bronchiectasis is defined as abnormal, chronic and permanent enlargement of one or more bronchi. Disease symptoms; often productive cough, dyspnea, fatigue and wheezing. Changing pulmonary mechanics, inadequate gas exchange, decreased muscle mass and associated psychological problems may cause dyspnea, decreased exercise capacity and health-related quality of life. Exercise training as a part of pulmonary rehabilitation is used to reduce the severity of symptoms; is an effective treatment to improve exercise capacity and health status. Virtual reality based exercise training has taken its place in many areas of rehabilitation as a current and new approach. In the studies in the literature, Nintendo Wii Fit games are an effective, motivating, entertaining and clinically useful method for reducing symptoms in the rehabilitation of chronic lung diseases. Wii Fit games generally include strengthening, aerobics and balance exercises. Developed by BreathingLabs, Breathing Games, which is based on breathing exercises, are a new product, a virtual reality application that has been included in a limited number of studies, has shown its effect on reducing respiratory problems and is open to research effects for many patient groups. The importance of this study is that it will be the first study on Nintendo Wii Fit games based exercise training and Breathing Games based breathing exercises training in children with bronchiectasis.

The aim of this study is to investigate the effect of different virtual reality-based exercise trainings on pulmonary function, respiratory and peripheral muscle strength, functional capacity and balance in children with bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Bronchiectasis diagnosis
* Stable clinical condition (no exacerbation in last 4 weeks)

Exclusion Criteria:

* Documented diagnosis of vestibular, neurological or orthopedic disorders which may affect balance and mobility
* Subjects previously involved in exercise training or physiotherapy programs
* Previous history of lung or liver transplantation

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2019-07-27 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-02-06 (Actual)

PRIMARY OUTCOMES:
Respiratory Function Test | Eight weeks
  Change from baseline Forced Vital Capacity (FVC) at 8 weeks
Respiratory Function Test | Eight weeks
  Change from baseline Forced Expiratory Volume in 1 second (FEV1) at 8 weeks
Respiratory Function Test | Eight weeks
  Change from baseline Peak Expiratory Flow (PEF) at 8 weeks
Respiratory Muscle Strength | Eight weeks
  Change from baseline maximum inspiratory pressure (MIP) at 8 weeks
Respiratory Muscle Strength | Eight weeks
  Change from baseline maximum expiratory pressure (MEP) at 8 weeks
Functional Capacity | Eight weeks
  Change from baseline distance covered in six-minute walk test at 8 weeks
Balance | Eight weeks
  Change from baseline postural stability test score in Biodex Balance System SD at 8 weeks
Balance | Eight weeks
  Change from baseline limits of stability test score in Biodex Balance System SD at 8 weeks
Balance | Eight weeks
  Change from baseline sensory integriation and balance test score in Biodex Balance System SD at 8 weeks
Peripheral Muscle Strength | Eight weeks
  Change from baseline M. Quadriceps strength at 8 weeks
Peripheral Muscle Strength | Eight weeks
  Change from baseline M. Biceps strength at 8 weeks
Peripheral Muscle Strength | Eight weeks
  Change from baseline handgrip strength at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif Universitesi, Department of Physiotherapy and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided